CLINICAL TRIAL: NCT05287620
Title: Objective, Passive Assessment of LRRK2 Carriers
Acronym: OPAL
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Emerald Innovations (Unknown); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Ray Dorsey, Professor, University of Rochester
Other Study IDs: STUDY00006771
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Emerald device — The Emerald device is a wireless sensor that can track the motion, breathing, and sleep of participants without touching or requiring any interaction with the participants, allowing them to go about their normal lives. The Emerald device operates by transmitting and receiving low power radio signals that reflect off of the participant and return back to the device. The power of these signals is 1,000 times lower than what a typical Wi-Fi device transmits. The ability of the device to monitor gait, breathing, sleep, and other metrics has been validated and documented. Studies of the Emerald device in individuals with Parkinson's disease, Alzheimer's disease, and rare diseases have demonstrated the feasibility of monitoring at home and the ability to characterize gait, breathing, and sleep in these populations specifically. In this study, the Emerald device will be used to characterize the mobility, breathing and sleep of the participant.

SUMMARY:
The goal of this project is to identify objective, sensitive, and convenient measures for assessing early signs of Parkinson's disease in an at-risk population at home. We will do so by using a wireless sensor and analyzing the radio signals that bounce off patients' bodies, while patients go about their normal life without needing to wear sensors, answer questionnaires, or actively perform any tests.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age
* Able and willing to provide informed consent
* English fluency
* U.S. resident
* LRRK2 G2019S gene carrier, determined by participation in VALOR-PD
* Mild parkinsonian signs, determined by modified Movement Disorder Society-Unifeid Parkinson's Disease Rating Scale (MDS-UPDRS) score from the most recent VALOR-PD visit
* Have WiFi in their residence
* Access to a smartphone or tablet

Exclusion Criteria:

* Inability to complete study activities, as determined by the study team
* Any medical or psychiatric condition that, in the study team's judgement, would preclude participation
* Self-reported or VALOR-PD investigator determined Parkinson's disease
* Any movement disorder (e.g. essential tremor)
* Currently taking neuroleptics or other drugs known to cause parkinsonism
* Pregnancy
* Non-ambulatory status
* More than one ambulatory pet in the household*
* More than two individuals in the household (not including participant)*

  * these criteria can be waived at the discretion of the investigators

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll LRRK2 G2019S carriers without self-reported or clinician-determined Parkinson's disease (PD) from the VALOR-PD study. VALOR-PD is an observational study following and characterizing a remote, nationwide cohort of LRRK2 G2019S carriers with (n = 59) and without PD (n = 218). Individuals who have a diagnosis of PD will not be eligible to participate, since we aim to explore the device's sensitivity in detecting early symptoms/signs of PD.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Gait speed | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ray Dorsey, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States